CLINICAL TRIAL: NCT06825143
Title: Therapeutic Strategies to Reduce Endothelial Ischemia-reperfusion Injury with Metabolic Syndrome: a Combination Approach with Lactate Administration and Ischemic Preconditioning
Brief Title: Therapeutic Strategies to Reduce Endothelial Ischemia-reperfusion Injury
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Gary Van Guilder (Other)
Responsible Party: Sponsor-Investigator, Gary Van Guilder, Principal Investigator, Western Colorado University
Organization: Western Colorado University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HRC-2024-02-06-R33
Record Dates: First submitted 2025-01-21; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Metabolic Syndrome; Vascular Injury; Ischemic Preconditioning; Endothelial Function (reactive Hyperemia); Endothelial Dysfunction
Keywords: endothelial ischemia/reperfusion injury; remote ischemic preconditioning; lactate; metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome; Vascular System Injuries; Hyperemia; Reperfusion Injury | interventions — Ischemic Preconditioning

STUDY DESIGN:
Intervention Model Description: The overall interventional study model will utilize a parallel design equivalence trial and a parallel design superiority trial. Both trials will have two Arms.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ischemic preconditioning versus intravenous lactate infusion (Active Comparator): To goal of this Arm is to compare the capacity of ischemic preconditioning (IPC) to protect against endothelial ischemia/reperfusion injury to the capacity of an intravenous lactate infusion to protect against endothelial ischemia/reperfusion injury. To achieve this goal, investigators will test the hypothesis that the capacity for intravenous lactate to reduce endothelial injury will be equivalent to that of IPC. Participants will be randomized to one of two Interventions. One Intervention will be the IPC intervention which is thought to be effective in treating the condition under study. The other intervention is the intravenous lactate intervention, which is the main focus of the study.
  Interventions: Procedure: Ischemic preconditioning; Drug: Intravenous lactate infusion; Procedure: No ischemic preconditioning (control); Drug: Normal Saline Infusion (Placebo)
- Ischemic preconditioning combined with an intravenous lactate infusion (Experimental): To goal of this Arm is to compare the capacity of ischemic preconditioning (IPC) combined with an intravenous lactate infusion to protect against endothelial ischemia/reperfusion injury to IPC by itself. To achieve this goal, investigators will test the hypothesis that the capacity to protect against endothelial injury will be better when IPC and lactate are combined compared to IPC alone. Participants will be randomized to one of two Interventions. One Intervention will be the IPC intervention by itself. The other intervention will be adding an intravenous lactate infusion together with IPC which is the main focus of the study.
  Interventions: Procedure: Ischemic preconditioning; Combination Product: Ischemic preconditioning and intravenous lactate

INTERVENTIONS:
Procedure: Ischemic preconditioning — The objective of this Intervention is to show that ischemic preconditioning (IPC) protects against endothelial ischemia/reperfusion injury. Baseline endothelium-dependent vasodilation to reactive hyperemia will be performed on the nondominant arm, followed by 3 × 5-minute cycles of IPC in the opposite arm. IPC will be induced using a blood pressure cuff placed on the opposite upper arm and inflated to 220 mmHg for 5 min, followed by 5 min of deflation. This procedure will be repeated two additional times taking about 30 minutest to complete. Following a 10-minute rest phase, endothelial injury will be induced using a blood pressure cuff that will be inflated to stop blood flow through the nondominant arm for 20 minutes, followed by 15 minutes of cuff deflation. Endothelium-dependent vasodilation measurements will be repeated immediately after the 15-minute cuff deflation phase.
Drug: Intravenous lactate infusion — The objective of this Intervention is to show that an intravenous infusion of lactate protects against endothelial ischemia/reperfusion injury. Baseline endothelium-dependent vasodilation to reactive hyperemia will be performed on the nondominant arm. Thereafter, a continuous intravenous infusion of lactate will be delivered in the contralateral arm. After systemic lactate reaches ~3 mmol/L, endothelial injury will be induced using a blood pressure cuff that will be inflated to stop blood flow through the nondominant arm for 20 minutes, followed by 15 minutes of cuff deflation. Endothelium-dependent vasodilation measurements will be repeated immediately after the 15-minute cuff deflation phase.
  Arms: Ischemic preconditioning versus intravenous lactate infusion
Procedure: No ischemic preconditioning (control) — The objective of this Intervention is to show that a control experiment without ischemic preconditioning does not provide protection against endothelial ischemia/reperfusion injury. Baseline endothelium-dependent vasodilation to reactive hyperemia will be performed on the nondominant arm, followed by 3 × 5-minute cycles of no upper arm occlusion in the opposite arm. To avoid upper arm occlusion, a blood pressure cuff will be placed on the upper arm and inflated to a low pressure of 20 mmHg pressure to not influence blood flow through the arm. This control procedure will be repeated two additional times taking about 30 minutes to complete. Following a 10-minute rest phase, endothelial injury will be induced using a blood pressure cuff that will be inflated to stop blood flow through the nondominant arm for 20 minutes, followed by 15 minutes of cuff deflation. Endothelium-dependent vasodilation measurements will be repeated immediately after the 15-minute cuff deflation phase.
  Arms: Ischemic preconditioning versus intravenous lactate infusion
Drug: Normal Saline Infusion (Placebo) — The objective of this Intervention is to show that a placebo intravenous infusion does not protect against endothelial ischemia/reperfusion injury. Baseline endothelium-dependent vasodilation to reactive hyperemia will be performed on the nondominant arm. Thereafter, a continuous infusion of normal saline that does not contain lactate will be delivered in the contralateral arm. After 20 minutes of the placebo infusion, endothelial injury will be induced using a blood pressure cuff that will be inflated to stop blood flow through the nondominant arm for 20 minutes, followed by 15 minutes of cuff deflation. Endothelium-dependent vasodilation measurements will be repeated immediately after the 15-minute cuff deflation phase.
  Arms: Ischemic preconditioning versus intravenous lactate infusion
Combination Product: Ischemic preconditioning and intravenous lactate — The objective of this Intervention is to show that combining ischemic preconditioning (IPC) with an intravenous infusion of lactate provides the best protection against endothelial injury. First, baseline endothelial function to reactive hyperemia will be performed on the nondominant arm. Thereafter, a continuous intravenous infusion of lactate will be delivered in the contralateral arm. After that investigators will administer IPC using a blood pressure cuff placed on the same upper arm and inflated to 220 mmHg for 5 min, followed by 5 min of deflation. This procedure will be repeated two more times taking about 30 minutes to complete. The intravenous lactate infusion will be maintained. After a 10-minute rest phase and while lactate is still being infused, endothelial injury will be induced using a blood pressure cuff inflated to stop blood flow through the opposite arm (nondominant arm) for 20 minutes, followed by 15 minutes of cuff deflation. Endothelial function will be repeated.
  Arms: Ischemic preconditioning combined with an intravenous lactate infusion

SUMMARY:
The objective of this clinical trial is to better understand how lactate, a naturally occurring energy substance, can be used to lessen damage to the vascular system in adults with a high cardiovascular disease risk.

The main questions it aims to answer are:

1. Does giving lactate intravenously reduce injury to the vascular system?
2. Does giving lactate intravenously together with blood flow occlusion - known as ischemic preconditioning, reduce vascular injury better than blood flow occlusion by itself?
3. How does lactate help the vascular system?

Researchers will compare lactate to a placebo (a look-alike substance that contains no lactate) to see if lactate works to lessen vascular injury.

Researchers will also compare lactate to blood flow occlusion to see which one is better at preventing vascular injury.

Researchers will also compare lactate and blood flow occlusion together to see if combining them works better than either one alone.

In one visit to the laboratory, participants will:

Obtain a measurement of vascular health in an arm Be given liquid lactate, a liquid placebo, and/or arm blood flow occlusion Obtain a second measurement of vascular health in an arm.

DETAILED DESCRIPTION:
Much of the mortality burden of ischemic heart disease is due to untreatable complications of ischemia-reperfusion (I/R) injury, greatly undermining the translation of cardioprotective interventions. Endothelial damage and dysfunction are centrally involved in many of the clinical consequences of myocardial I/R injury. While a very promising therapeutic defense mechanism against I/R-induced endothelial dysfunction is ischemic preconditioning (IPC), it has not fared well in multi-center phase III clinical trials. Complementary strategies that elicit additive or synergistic benefits against I/R injury are urgently needed. Because lactate has extensive endothelial protective effects, the recruitment of additional protective pathways with lactate that cannot be activated with IPC alone provides an innovative and powerful strategy to greatly enhance cardioprotection in the clinical arena. Little is understood about whether including lactate with IPC as a dual approach can bolster protection in adults with CVD risk in which the endothelial protective effects of IPC are already weakened. The long-term goal of this research is to develop improved combination therapeutic strategies to expedite the clinical application of IPC for cardioprotective purposes. The objective is to better understand how lactate administration can be used to alleviate endothelial I/R injury. In a model of endothelial I/R injury, our central hypothesis is that lactate administration alone will reduce endothelial dysfunction, and when included as a combination strategy with IPC, will improve protection with metabolic syndrome. The rationale for the proposed research is based on the poor translatability of existing cardioprotective strategies to date. The central hypothesis will be tested by pursuing three aims: 1) Determine the degree to which lactate administration attenuates endothelial I/R injury; 2) Determine the superiority of a combined multi-targeted therapeutic strategy against endothelial I/R injury in adults with metabolic syndrome; and 3) Establish mechanistic insight into the endothelial protective effects of lactate. In Aim #1, the investigators will utilize a randomized equivalence trial comparing the effects of lactate administration versus IPC on endothelial function in 32 adults. For Aim #2, a randomized superiority trial in 36 adults with metabolic syndrome will compare the dual effects of IPC combined with lactate versus IPC alone. For Aim #3, a series of biomarker studies by which lactate is likely to modify the therapeutic response to I/R injury are proposed. For Aims #1 and #2, endothelium-dependent vasodilation (primary endpoint) will be compared between trials for equivalence, and superiority, respectively. For Aim #3, the investigators expect lactate will protect against endothelial I/R injury, in part, by reducing circulating microparticles of endothelial activation and vascular inflammation, and increasing total antioxidant capacity, nitric oxide bioavailability, and angiogenic factors. The approach is conceptually innovative because the findings are likely to be the first in vivo evidence supporting the development of a multi-faceted approach that exploits the potential for synergistic cytoprotection involving IPC combined with lactate. This contribution would advance the development of new translatable strategies for cardioprotection.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary men and women between the ages of 18-65 years of all races and ethnicity
* Diet and weight stable for the past 3 months
* Non-smoking and not using tobacco or electronic cigarettes

Exclusion Criteria:

* Use of medications known to affect cardiovascular function
* Hyperlactemia
* Type A lactic acidosis
* Type B lactic acidosis
* Extracellular hyperhydration or hypervolemia
* Hyperkaliemia
* Hypercalcemia
* Metabolic alkalosis
* Metabolic acidosis
* McArdle's Disease
* Diabetes Type 1 and 2
* Taking oral contraceptives or hormone replacement therapy
* Body mass index greater than or equal to 35
* Smoking or using smokeless tobacco and electronic cigarettes
* Cardiovascular, cerebrovascular, liver, respiratory, and renal disease
* Atrial fibrillation or other sustained supraventricular/ventricular arrhythmia
* Familial hypercholesterolemia
* Rheumatoid arthritis
* Sleep apnea
* Currently pregnant, recent pregnancy, or breast-feeding
* Autonomic nervous system dysfunction
* Raynaud's disease
* Active malignancy excluding basal cell carcinoma of the skin
* Three or more days of at least 30 minutes of aerobic exercise in the past 3 months
* Inability to provide consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Baseline value of the mean peak forearm blood flow response to reactive hyperemia. | Baseline (time 0)
  Endothelium-dependent vasodilation will be assessed in the experimental (nondominant) arm by the forearm blood flow response to reactive hyperemia using strain-gauge venous occlusion plethysmography. Data are reported in ml of blood per 100 mL arm volume per minute.
Mean peak forearm blood flow response to reactive hyperemia at 3 hours. | At 3 hours
  Endothelium-dependent vasodilation will be assessed in the experimental (nondominant) arm by the forearm blood flow response to reactive hyperemia using strain-gauge venous occlusion plethysmography. Data are reported in ml of blood per 100 mL arm volume per minute.

CONTACTS AND LOCATIONS:
Locations (1):
- High Altitude Physiology Laboratory at Western Colorado University, Gunnison, Colorado, United States

IPD SHARING:
Plan to Share IPD: No